CLINICAL TRIAL: NCT01972971
Title: To Establish a Novel Prototype of Clinical Pharmacy Services by Warfarin Consultation in a Pharmacist Clinic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 201105109RC
Record Dates: First submitted 2013-10-13; First posted 2013-10-31 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Intentional Warfarin Sodium Overdose
Keywords: warfarin; pharmacist; anticoagulation
MeSH Terms: interventions — Patient Education as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pharmacist care (Other)
  Interventions: Other: patient education

INTERVENTIONS:
Other: patient education — one by one patient education

SUMMARY:
Warfarin, the major oral anticoagulant currently available in Taiwan, is used for the prevention and treatment of a variety of thromboembolic disorders. Under dosing of warfarin may cause treatment failure and over dosing may cause bleeding because of its narrow therapeutic index. Therefore, it is important to monitor prothrombin time (PT) and international normalize ratio (INR) periodically in order to evaluate the appropriateness of warfarin dosing.

Lots of factors influencing warfarin anticoagulation effects include polymorphisms of Cytochrome P450 2C9(CYP2C9)and Vitamin K epoxide reductase complex subunit 1(VKORC1)genes, age, weight, diet and concurrent medications. Taking into consideration of physicians' work load, pharmacist-managed anticoagulation clinics were set up to help strengthen patient care in US to ensure patient medication safety. In addition, differences in genetic polymorphisms between Chinese and Caucasian have great impacts on warfarin dosage, and there is still no consensus on warfarin utilization guideline in Taiwan. Pharmacist-managed anticoagulation clinics provide individualized care, consistent monitoring and patient education. Through this service, physicians can get the latest integrated information about their patients, patients themselves are more familiar with their medication, and adherence can be improved. Therefore, those who take warfarin will get better INR control, less adverse drug-related events and treatment failure.

This is the first prototype of pharmacist clinic for a specific medication in our hospital. The adverse drug events and coagulation function data collected through this program can be used for the implementation of warfarin treatment guideline in Taiwan in the future. The impact of pharmacist clinic can be evaluated by questionnaire of satisfaction and knowledge survey. It can be used as a model for implementing other pharmacist-managed clinics and improving patient medication safety.

ELIGIBILITY:
Inclusion Criteria:

* >20 y/o
* Has been received warfarin therapy for 3 months and anticipated treatment duration of more than 3 months and a week
* Has legitimate indication for warfarin
* Has the capacity to understand the condition and implications of anticoagulant therapy

Exclusion Criteria:

* Who can't be regular follow-up at National Taiwan University Hospital.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2012-02; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
percentage of INR in therapeutic range and incidence of complications | 3 months
  The INR value collected during the 3 months before enrollment and within 3 months after enrollment, which was proceeded by the one month wash-out period. The bleeding or thromboembolic events during this period were also collected. The outcome was assessed by the percentage of patient time with INR within the target range (1.8-2.4) and incidence of complications.

SECONDARY OUTCOMES:
patient's warfarin knowledge improvement | 3 months
  Patient's warfarin-related knowledge would be assessed by questionnaire. The validity of the questionnaire were assessed by experts. This questionnaire contained 9 aspects. the pre-test of warfarin-related knowledge questionnaire was conducted before patient education, and the post-test was conducted 2 months after enrollment in the pharmacist clinic. The correct percentage between pre-test and post-test would be compared.
Patient's satisfaction to anticoagulation pharmacist clinic | 3 months
  Patient's satisfaction would be assessed by questionnaire. The validity of the questionnaire was assessed by experts. The per-test was conducted before the patient enrolled to pharmacist clinic, and the post-test was conducted 2 months after enrollment. The difference between pre-test and post-test would be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Fe-Lin L WU, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan